CLINICAL TRIAL: NCT02233556
Title: Effects of Memantine on Event-related Potential in the Comparison of Patients With Early Schizophrenia and Healthy Subjects
Brief Title: Effect of Memantine on ERP in Early Schizophrenia and Healthy Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 201308083MINB
Record Dates: First submitted 2014-02-26; First posted 2014-09-08 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Schizophrenia
Keywords: event-related potential; mismatch negativity; NMDA; Glutamate
MeSH Terms: conditions — Schizophrenia | interventions — Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Memantine (Experimental): This study has only one arm. i.e. Single dose of memantine 20mg
  Interventions: Drug: Memantine

INTERVENTIONS:
Drug: Memantine — Taking 20mg(2 capsules) of memantine, followed by Event related potential assessments as below:
  1. Mismatch negativity(MMN)
  2. P50
  Other Names: Ebixa 10 mg, manufactured by Lunbeck A/S, Denmark

SUMMARY:
Patients with schizophrenia are deeply affected by the positive symptoms, negative symptoms and cognitive impairment. A generalized cognitive deficit could be frequently observed and traced back to early stage of the disease. Currently medication intervention significantly improves positive symptoms through dopamine receptor modification, leaving alone the negative symptoms and cognitive impairment. Besides dopamine dysregulation, more and more attention had been paid to the association of N-methyl-D-aspartate (NMDA) type glutamate receptor and schizophrenia, focusing on the neurobiological and cognitive biomarkers change. Memantine, an uncompetitive antagonist of NMDA type glutamate receptor approved as cognitive enhancer for Alzheimer's disease, is a potential candidate for preventing cognitive decline of schizophrenia. Previous randomized clinical trials failed to demonstrate its efficacy on chronic schizophrenic patients and it might be related to the chronic and irreversible disease process. There is also study supporting that memantine induces change in mismatch negativity (MMN) in frontal cortex of healthy subjects. This study will compare the MMN change of healthy subjects and the population of early schizophrenia, who has persistent neurobiological, cognitive biomarkers or negative symptoms despite subsided positive symptoms. Both male and female aged 20-45 years old outpatients with a length of illness for less than 5 years since first diagnosed as schizophrenia, currently receiving treatment by atypical antipsychotics in a relatively stable condition will be recruited. Healthy subjects will be recruited comparing their age and sex. We plan to recruit 10 subjects for both patient and healthy subjects with a total of 20 participants. All participants will receive general clinical, cognitive and event-related potential (ERP) evaluation as baseline before taking medication. Twenty mg of memantine will be given 4 hours before ERP retest. The analyses will be performed based on the change of ERP using paired-t sample test. Baseline clinical and cognitive symptoms will be analyzed as possible confounders.

DETAILED DESCRIPTION:
In this proposal, we use one-dose memantine trial to compare the difference of MMN change between healthy subjects and early schizophrenia patients. The cognitive and negative symptoms will be counted as possible confounding variables. We would like to make connection and association between neurobiological and neurocognitive markers for further treatment application.

The specific aim of this project is to test if memantine will influence the ERPs change, as in healthy subjects, in patients with early schizophrenia. The specific study population is been known of just have their first episode psychosis subsided, conventionally defined by significantly improved positive symptoms, yet some of them complaining of cognitive decline or presenting with persistent negative symptoms. Previous study showed improvement in mismatch negativity was correlated with general function improvement in schizophrenia. Although a recent study failed to demonstrate positive effects on residual psychopathology of a group of chronic stable schizophrenic patients. In this study we are targeting at a specific population of early schizophrenic patients to examine the efficacy of memantine on neurobiological markers and possible application to general psychopathology. Our objectives include:

1. Test memantine effects on the change of ERPs, especially focus on mismatch negativity.
2. Compare the ERP difference between healthy subjects and early schizophrenic patients
3. Examine whether the effect of memantine will be affected by any significant baseline clinical variables or predisposed cognitive deficits.

First if we could replicate the ERP change in healthy subjects influenced by memantine, and we could further compare the difference between healthy subjects and patient subjects. It may support the hypothesis of NMDA-type glutamate receptor dysregulation theory in schizophrenia. If further association is detected through larger scale study between ERP and clinical symptoms, we could apply memantine in the add-on treatment of schizophrenia. As memantine is already an approved medicine for treatment of moderate to severe Alzheimer disease in many countries worldwide, hopefully we can add a new indication to its original clinical application. Thus it will become the first medicine that can help a condition which has rendered a lot of schizophrenic patients marked impairments in their social and occupational functioning from the early stage of their life. We believe this impact will be even bigger than the original indication of memantine, which is exclusively for patients with dementia. Rather than delaying deterioration of cognitive functioning in patient's late life, an adjuvant therapy for early intervention in schizophrenia aiming at improving cognitive function and hence restoring social and occupational functioning bears greater impact on a patient's life trajectory and lessen the burden of a society. Furthermore, the results from this project will provide critical evidence to support or refute the hypoglutaminergic theory of schizophrenia, which might be an important complement to the hyperdopaminergic theory. With a better understanding of the pathophysiology of schizophrenia not only focusing on dopaminergic system-related positive symptoms but also glutamatergic system-related cognitive and negative symptoms, will provide theoretic base of psychopharmacology in developing agents targeting at different systems to improve the outcome of schizophrenia from the early stage or even the putative pre-psychotic stage of the illness.

ELIGIBILITY:
Inclusion criteria for patient subjects:

1. Both male and female outpatients
2. Age 20-45 years old at the time of screening
3. A diagnosis of schizophrenia based on the Structured Clinical Interview for DSM-IV
4. A duration of illness for less than 5 years since initially diagnosed as schizophrenia
5. Currently receiving treatment mainly by an atypical antipsychotic (risperidone, olanzapine, amisulpiride, aripiprazole, quetiapine, ziprasidone, paliperidone), including long-acting injectable antipsychotic
6. A first generation antipsychotic agent only for a low-dose, as needed use purpose
7. No revised use of benzodiazepines, antidepressants, anticholinergics, or other concomitant medications during past 3 months

Inclusion criteria for healthy subjects:

1. Both male and female
2. Age 20-45 years old at the time of screening
3. No psychiatric diagnosis based on the Structured Clinical Interview for DSM-IV
4. No current use of any pharmaceutical agents in past 2 weeks

Exclusion criteria for all participants:

1. A score of 5 or more on any of the 7 positive symptom items of the PANSS rating at screening
2. Scores of 4 on at least 3 of the 7 positive symptom items of the PANSS rating at screening
3. A major relapse resulting in readmission or doubling the dosage of previous effective antipsychotic treatment during the course of illness
4. A change of current antipsychotic medication in recent 3 months
5. Mental retardation known as IQ below 70 prior to the diagnosis of schizophrenia
6. A history of pervasive mental disorder or bipolar disorder
7. A medical condition with significant cognitive sequelae
8. A history of substance dependence
9. A history of hypersensitivity to memantine or other drugs of the same class, such as amantadine
10. Pregnancy, plan to get pregnant during the study period, or lactating women
11. Abnormal liver function (AST, ALT higher than doubling the upper limits of normal range) or abnormal renal function (blood creatinine > 1.3 mg/dL)
12. A history of epilepsy
13. A history of myocardial infarction, congestive heart failure, uncontrolled hypertension, stroke, or severe heart block.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Changes in auditory event-related potentials "MMN"before/after intake of a single dose memantine | 4 hours after intake of a single dose memantine
  Previous studies revealed deficits in cognition via auditory event-related potential, such as Mismatch Negativity. This study would compare the effect of single dose memantine in MMN.

SECONDARY OUTCOMES:
Changes in auditory event-related potentials "P50" before/after intake of a single dose memantine | 4 hours after intake of a single dose memantine
  Previous studies revealed deficits in cognition via auditory event-related potential, such as P50. This study would compare the effect of single dose memantine in P50

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Hsien Hsieh, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan